CLINICAL TRIAL: NCT02811640
Title: Development of a Simplified Method to Measure Intra-abdominal Pressure in Peritoneal Dialysis Patients
Brief Title: Intra-abdominal Pressure in Peritoneal Dialysis Patients
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 20160377-01H
Record Dates: First submitted 2016-06-21; First posted 2016-06-23 (Estimated); Results first posted 2020-11-18 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-10

CONDITIONS: Peritoneal Dialysis
Keywords: Intra-Abdominal Pressure; Stryker Pressure Monitor
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study Participants: Adults with chronic kidney disease who will have a PD catheter inserted at the Ottawa Hospital
  Interventions: Other: Study Participants

INTERVENTIONS:
Other: Study Participants — IAP will be observed and measured with a hand held Stryker Pressure Monitor during laparoscopic surgery and compared to the standard IAP measurements obtained with the insufflator at the time of PD catheter insertion
  Other Names: Observation

SUMMARY:
Patients treated with peritoneal dialysis (PD) are at increased risk of developing mechanical complications such as dialysate leaks and hernias thought to be related to an increase in intra-abdominal pressure (IAP) secondary to the addition of dialysate to the abdomen. Resistance training has been shown to increase IAP but it is unclear in the general population and in patients treated with PD if this training increases the risk of developing hernias.

This study is observing the difference in IAP pressure measurements obtained by the Stryker intracompartmental (STIC) pressure monitor versus the standard IAP pressure measurements obtained with the insufflator at the time of PD catheter insertion.

DETAILED DESCRIPTION:
Ten patients who are having a peritoneal dialysis (PD) catheter inserted at the Ottawa Hospital, and who provide informed consent, will undergo intra-abdominal pressure (IAP) measurements with the Stryker intracompartmental (STIC) pressure monitor. Values will be compared to the insufflator at inflation pressures 5,10, and 15 mmHg (millimeters of mercury).

To determine if the Stryker pressure monitor is appropriate for measuring IAP in PD patients, the observed pressures will be analyzed with Bland Altman plots. If the mean difference between readings is 5 mmHg and 95% of the points fall within 2 standard deviations of the mean difference, the Stryker pressure monitor will be considered an acceptable method of measuring IAP.

This tool will then be used as part of a future larger trial which will 1) measure IAP with resistance training in patients treated with PD; with and without dialysate, 2) assess PD patient interest in participating in resistance training trials and 3) determine the appropriateness of the proposed resistance training program for this patient population.

The ultimate goal is to use this study to help inform and develop a clinical trial to 1) assess the impact of resistance training on quality of life and functional status, 2) assess the risk of developing leaks/hernias, and 3) determine if there is an association between IAP during resistance training and subsequent hernia development

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years old)
* Chronic kidney disease
* Will have a PD catheter inserted in the operating room at the Ottawa Hospital using laparoscopic surgery

Exclusion Criteria:

* Patients who will have a non-standard PD catheter insertion position (eg parasternal)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (>18 years old) with chronic kidney disease that will have a PD catheter inserted in the operating room at the Ottawa Hospital using laparoscopic surgery
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2016-06-30 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2019-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Zimmerman, MD, MSc, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two patients had to be excluded from the analysis due to difficulties zeroing the Stryker pressure monitor at the time of surgery.
Period: Overall Study
Arm/Group | Study Participants
Started | 12
Completed | 10
Not Completed | 2
Not completed — Technology malfunction | 2

BASELINE CHARACTERISTICS:
Arm/Group | Study Participants
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 12

OUTCOME MEASURES:

1. Primary Outcome: Intra-Abdominal Pressure (IAP)
Description: The Intra-Abdominal Pressure (IAP) measured with the Stryker monitor connected to the peritoneal dialysis (PD) catheter was compared with the insufflator pressures at of 15, 10, and 5 mm Hg.
Time Frame: During laparoscopic surgery, up to 30 minutes
Population: There is only 1 arm or group for this study. The study participants are adults with chronic kidney disease who had a PD catheter inserted at the Ottawa Hospital. During the insertion, IAP was observed and measured with a hand held Stryker Pressure Monitor and with the insufflator. These results were compared, and the average difference and the standard deviation between the two are reported.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Study Participants
Number analyzed (Participants) | 10
mm Hg
  15 mm Hg | -0.5 (2.0)
  10 mm Hg | -0.2 (3.1)
  5 mm Hg | -1.2 (2.6)

ADVERSE EVENTS:
Time Frame: During laparoscopic surgery, up to 30 minutes
Arm/Group | Study Participants
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

LIMITATIONS AND CAVEATS:
Technical problems with measurement leading to small sample size, and lack of a gold standard comparative may have affected our results.

.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-25): https://cdn.clinicaltrials.gov/large-docs/40/NCT02811640/Prot_SAP_000.pdf